CLINICAL TRIAL: NCT05629442
Title: A Study of the Role of Circulating Tumor DNA in Predicting the Likelihood of Organ Preservation or Pathologic Complete Response After Neoadjuvant Therapy for Rectal Cancer
Brief Title: ctDNA and Organ Preservation/Pathologic CR in Rectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: C2i Genomics (Industry); Spier Family Foundation (Unknown)
Responsible Party: Principal Investigator, Theodore Sunki Hong, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 22-244
Record Dates: First submitted 2022-09-14; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Rectal Cancer; Non Metastatic Rectal Cancer
Keywords: Rectal Cancer; Non Metastatic Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biospecimen submission should include both tissue and blood samples:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EVALUATION OF CTDNA: This prospective observational, non-therapeutic study will enroll patients with T3, T4, or node positive rectal cancer eligible to undergo total neoadjuvant therapy/ All procedures involved with this trial will be done as per standard of care
  - Except for the initial research biopsy, quality of life assessments and ctDNA collection
  Interventions: Other: ctDNA

INTERVENTIONS:
Other: ctDNA — initial research biopsy, quality of life assessments and ctDNA collection

SUMMARY:
This prospective observational, non-therapeutic study for patients with T3, T4, or node positive rectal cancer eligible to undergo total neoadjuvant therapy.

This research study involves the collection of data and biospecimens (blood and tissue) to see if the presence of circulating tumor DNA (genetic material) ctDNA will help monitor rectal cancer more closely and potentially detect a recurrence before routine scans, performed per standard of care

C2i Genomics, a biotechnology company, and the Spier Foundation are supporting this research study by providing funding for the study.

DETAILED DESCRIPTION:
The research study procedures include screening for eligibility and the collection of data and biospecimens. Non-operative management is offered as part of routine clinical care.

It is expected that up to 60 participants will be enrolled, with the goal that 55 participants will take part in this research study .

Participants enrolled on the study will remain on study for up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants with T3, T4, or node-positive non-metastatic rectal cancer.
* Participants must have original tumor tissue (formalin-fixed, paraffin embedded specimens) available for analysis or be willing to undergo a baseline research biopsy.
* Participants must be 18 years of age or older.
* ECOG 0-2.
* Participants must be eligible for at least 3 months of FOLFOX, FOLFIRINOX/FOLFOXIRI, or CAPOX
* Participants must be eligible for long course chemoradiation to 40-54 Gy.
* Participants must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

* Participants must not have any other organ cancer evident at the time of enrollment.
* Participants may not have any other concurrent serious illness that makes participation on this study impractical or clinically inappropriate.
* Participants must not be actively or planning to be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective observational, non-therapeutic study will enroll patients with T3, T4, or node positive rectal cancer eligible to undergo total neoadjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Rate of successful non-operative management | 1 year
Rate of successful pathologic complete response | 1 year

SECONDARY OUTCOMES:
Rate of local recurrence | 5 years
  Local recurrence is defined as cancer coming back is in the same place as the original cancer or very close to it. Local recurrence will be assessed in participants who achieved a Clinical Complete Response (cCR) or Near Complete Clinical Response (nCR) after rectal cancer treatment by ctDNA status with the C2i assay.
EORTC-QLQ-CR 29 questionnaire | Up to 30 months
  European Organization for Research and Treatment of Cancer-Colorectal surgery (EORTC-QLQ-CR 29) is a 29-item patient-reported questionnaire to assess health-related quality of life in patients with colorectal cancer.
  Each question ranges in score from 1 to 4. Higher scores indicate higher levels of symptoms or less functioning.
FACT-C questionnaire | Up to 30 months
  Functional Assessment of Cancer Therapy- Colorectal (FACT-C) is a 37-item patient-reported questionnaire to assess quality of life in patients with colorectal. FACT-C questions are divided into four primary quality of life domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being.
  Participants rate each item on the questionnaire from 0 to 4. Total score range is from 0 to 136. Higher scores generally indicate better quality of life.
IADL Scale | Up to 30 months
  Instrumental Activities of Daily Living (IADL) Scale is an 8-item patient-reported questionnaire with a summary score from 0 (low function) to 8 (high function).
  IADLs are things you do every day to independently take care of yourself and your home.
Brief Pain Inventory (BPI) questionnaire | Up to 30 months
  Brief Pain Inventory (BPI) is a questionnaire to measure the severity and interference of pain on daily functions in participants with cancer.
  BPI scale total score:
  * worst pain score: 1-4 = mild pain
  * worst pain score: 5-6 = moderate pain
  * worst pain score: 7-10 = severe pain
Bowel function assessment with LARS score | Up to 30 months
  Low Anterior Resection Syndrome (LARS) score (LARS) is a 5-item questionnaire to assess bowel dysfunction following a low anterior resection for rectal cancer.
  LARS total score:
  * 0-20 = no dysfunction
  * 21-29 = minor dysfunction
  * 30-42 = major dysfunction
Bowel function assessment with FISI score | Up to 30 months
  Fecal Incontinence Severity Index (FISI) is a patient-reported questionnaire that helps quantify the impact of adult incontinence leakage on quality of life.
  Total score range is from 0 to 61. Higher scores indicate a higher perceived severity of fecal incontinence and related impact on quality of life.
Bowel function assessment with FIQOL score | Up to 30 months
  Fecal Incontinence Quality of Life (FIQOL) is a 29-item patient-reported questionnaire to assess quality of life of participants with fecal incontinence. The questionnaire has 4 subscales: lifestyle, coping/behavior, depression/self-perception and embarrassment.
  Subscale scores range from 1 to 5 and are the average response to all items on each scale. Total FIQOL score is the sum of all four subscales. Lower scores indicate lower functional status and related quality of life.
Disease-free survival (DFS) | Up to 30 months
  Disease-free survival (DFS) is defined as the length of time after completion of rectal cancer treatment that the patient survives without any signs or symptoms of that cancer.
Overall Survival (OS) | Up to 30 months
  Overall survival (OS) is defined as the length of time after starting rectal cancer treatment that participants are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore S. Hong, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mass General Cancer Center Newton-Wellesley Hospital, Newton, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation